CLINICAL TRIAL: NCT02249403
Title: Efficacy and Safety of 6, 12, 24, and 36 mg Tid po and 36 mg Bid po Talsaclidine (Free Base) for 12 Weeks in a Double-blind, Randomised, Placebo-controlled Parallel Group Comparison in Patients With Mild to Moderate Dementia of Alzheimer Type
Brief Title: Efficacy and Safety of Talsaclidine in Patients With Mild to Moderate Dementia of Alzheimer Type
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 506.203
Record Dates: First submitted 2014-09-23; First posted 2014-09-25 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

ARMS (6):
- Talsaclidine, 6 mg tid (Experimental)
  Interventions: Drug: Talsaclidine 6 mg
- Talsaclidine, 12 mg tid (Experimental)
  Interventions: Drug: Talsaclidine 12 mg
- Talsaclidine, 24 mg tid (Experimental)
  Interventions: Drug: Talsaclidine 24 mg
- Talsaclidine, 36 mg tid (Experimental)
  Interventions: Drug: Talsaclidine 36 mg
- Talsaclidine, 36 mg bid (Experimental)
  Interventions: Drug: Talsaclidine 36 mg; Drug: Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Talsaclidine 6 mg
  Arms: Talsaclidine, 6 mg tid
Drug: Talsaclidine 12 mg
  Arms: Talsaclidine, 12 mg tid
Drug: Talsaclidine 24 mg
  Arms: Talsaclidine, 24 mg tid
Drug: Talsaclidine 36 mg
  Arms: Talsaclidine, 36 mg bid; Talsaclidine, 36 mg tid
Drug: Placebo
  Arms: Placebo; Talsaclidine, 36 mg bid

SUMMARY:
The objective of this trial was to assess the dose-response relationship of symptomatic efficacy of talsaclidine base on ADAScog and to assess safety and tolerability

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient, age: over 40 years (lower age if genetic Dementia of Alzheimer Type (DAT) is documented. Patients over 85 years need to be in a clinically stable state (investigator's judgement)
* Patient's educational level is > 4 years
* Patient is able to understand the patient information and give informed consent
* Patient has given written informed consent in accordance with Good Clinical Practice and local legislation
* Patient has a non-demented relative or care giver who is willing to support the clinical trial; his/her written informed consent is optional
* Body weight: within +/- 30% of normal weight (Broca index)
* Diagnosis of DAT by the National Institute of Neurological and communicative Disorders-Alzheimer's Disease and Related Disorder Association (NINCDS-ADRDA) criteria
* MMS-score 10 - 24 inclusive
* Rosen ischemia score is lower or equal to two
* Patient is able to complete the trial examinations, to hear, speak, read and write in a basic way and primary sensorial functions are intact

Exclusion Criteria:

* Any dementia of vascular genesis (excluded by Rosen ischemia score > 2)
* Magnetic Resonance Imaging (MRI) or Computer Tomogram (CT) (more recent than 12 months; if a MRI of CT recording is performed more than 12 months before study entry, it must be repeated) findings make the diagnosis of DAT unlikely
* Any stroke history
* All secondary dementia (exclusion diagnosis defined by the NINCDS-ADRDA criteria) as a late complication of:

  * Cranio-cerebral trauma
  * Intoxication (incl. history of alcohol and drug abuse)
  * Cerebral infections (e.g. neurosyphilis)
  * Thyroid dysfunction
* Cerebral dysfunction due to metabolic disorders (e.g. unstable thyroid dysfunction, or unstable insulin-dependent diabetes mellitus with hypo-/hyper-glycemic episodes)
* Deficiency of vitamin B12 or folic acid as a reason of dementia
* Brain tumour (A patient with an incidental tumour found on CT not felt to be clinically relevant may be included, i.e.: meningioma)
* Down's syndrome, Parkinsonism, Huntington's chorea
* Multiple sclerosis
* Major depression defined by the Hamilton Depression Rating Scale (HAMD) 17 item scale (≥ 16)
* Depressive pseudo dementia
* Mental retardation
* Hydrocephalus
* Epilepsy
* Endogenous psychoses (schizophrenia)
* Untreated or non-compensated hypertension (Blood Pressure systolic > 180 and/or diastolic > 110 mmHg)
* Hypertension being treated with reserpine, clonidine or β-blockers (these cases have to be adjusted to therapy with e.g. calcium antagonists 4 weeks before start of treatment)
* Severe heart failure (NYHA: III and IV)
* Arrhythmias (Lown: II-IV, Electrocardiogram > 30 ventricular extrasystoles/hour, multifocal or multiform and repetitive forms of ventricular extrasystoles)
* Bronchial asthma with phases of exacerbation or inducible by aspirin or other Nonsteroidal anti-inflammatory drugs
* Severe diabetes mellitus: insulin dependent and not stabilised (patient with an HbA1c in normal range, clinically stable diabetes and any case of insulin dose ≤ 0.5 UI/kg/day may be included), or other metabolic diseases
* Renal insufficiency: calculated creatinine clearance is less than 60 ml/min
* Acute hepatic disorder (liver enzymes above 50 % upper normal limit)
* Chronic hepatitis within the last two years (positive hepatitis titer, Hepatitis A Virus, Hepatitis B Virus, Hepatitis C Virus, cytomegalovirus, Epstein-Barr virus or abnormal immunological values (positive immunoglobulin M(IgM)/IgG) are allowed if all liver enzymes are within the normal range)
* Recent history of liver disease (2 years) including drug intoxication (e.g. narcotics, cytostatics etc.)
* Patients with obvious symptoms of dehydration
* History of drug or alcohol abuse or dependence on other hepatotoxic agents (if a patient is permanently hospitalised and a drug screen performed at the beginning of hospitalisation, no additional drug screen is necessary)
* Neoplasm currently active or likely to recur (except basal cell carcinoma)
* Participation in another clinical trial within the last four weeks and re-entering from this or a previous talsaclidine trial
* Pregnant and lactating woman, woman with childbearing potential not using an approved method of contraception
* Insufficient compliance: in the investigator's opinion the patient or family is unable to comply with the protocol requirements

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 1999-01; Primary Completion 2000-01 (Actual)

PRIMARY OUTCOMES:
Change in Alzheimer's Disease Assessment Scale cognitive part (ADAScog) | Baseline, week 12

SECONDARY OUTCOMES:
Change in ADAScog (extension) | Baseline, week 4, 8 and 12
  measures cognitive capability
Change in ADAScog (Total) | Baseline, week 4, 8 and 12
  Defined as ADAScog + ADAScog (Extension)
Change in mini mental state (MMS) | Screening, week 12
Change in neuropsychiatric inventory (NPI) | Baseline, week 12
  measures behavioural symptoms
Change in Hamilton Depression Rating Scale | Screening, week 12
  measures depressive mood
Change in instrumental activity of daily living (IADL) | Baseline, week 12
  measures functional performance
Change in living status rated on a 6-point verbal rating scale | Baseline, week 12
Change in clinician's global impression rated with Alzheimer's Disease cooperative Study - Clinical Global Impression of Change (ADCS-CGIC) | Baseline, week 12
Number of patients with adverse events | up to 12 months